CLINICAL TRIAL: NCT00789386
Title: The Effect of Remifentanil on Established Capsaicin-Induced Hyperalgesia in Human Volunteers
Acronym: RemiCaps2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Professor Burkhard Gustorff, Vienna Human Pain Research Group, Department of Anaesthesia, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: VHPRG-RemiCaps2; LS07-040
Record Dates: First submitted 2008-11-10; First posted 2008-11-11 (Estimated); Last update posted 2009-05-21 (Estimated); Status verified 2009-05

CONDITIONS: Hyperalgesia
Keywords: Capsaicin; Remifentanil; Hyperalgesia
MeSH Terms: conditions — Hyperalgesia | interventions — Remifentanil; Midazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Remifentanil (Experimental)
  Interventions: Drug: Remifentanil
- Midazolam (Placebo Comparator): Active Placebo
  Interventions: Drug: Midazolam

INTERVENTIONS:
Drug: Remifentanil — Remifentanil (Ultiva ®; Glaxo-Smith-Kline; Vienna, Austria) at an initial dose of 0.24 µg kg-1 min-1 will be applied iv during 60 minutes.
  Arms: Remifentanil
Drug: Midazolam — Midazolam (Dormicum®; Roche; Vienna, Austria) will be applied iv as active placebo at a dose of 7.5 µg.kg-1.min-1 over 10 minutes to mimic typical central nervous side effects of remifentanil.
  Arms: Midazolam

SUMMARY:
Treatment of chronic pain is a major clinical challenge since chronic pain is frequent and leads to deterioration of quality of life. An injury or wound can lead to long term changes in the nervous system that make the skin more sensitive at and near the injury; this is termed hyperalgesia and occurs through long term depotentiation (LTP), i.e., a change in the synaptic interaction between neurons.

Opioids are the gold standard for the symptomatic therapy of moderate to severe pain. Now, in animal studies the investigators have discovered previously unrecognized effects of opioids.

Intradermal injection of capsaicin (injection of pepper extract into the skin) is an established pain model in humans. The investigators want to test the influence of remifentanil, an ultra-short acting opioid, on hyperalgesia observed after intradermal capsaicin in human volunteers in a double blind cross-over prospective active placebo controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination
* Drug free for 1 week prior to the study day

Exclusion Criteria:

* Regular use of medication especially analgesics
* Abuse of alcoholic beverages, drug abuse
* History of asthma
* Participation in a clinical trial in the 2 weeks preceding the study
* Symptoms of a clinically relevant illness in the 2 weeks before the first study day
* Resting systolic blood pressure > 135 mmHg or diastolic blood pressure > 85 mmHg
* Acute skin diseases like sunburn on the relevant areas or skin lesions
* Pregnancy or breast feeding

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-10 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Area of pin prick hyperalgesia | 0-6 hours

SECONDARY OUTCOMES:
Stimulus-response (SR)function to a set of modified rigid von Frey filaments (8-512 mN) | 0-6 hours
Pain immediately after injection | 0-15 minutes
Heat pain threshold within the area of mechanical hyperalgesia | 0-6 hours
Mechanical pain threshold within the area of pin prick hyperalgesia, area of dynamic allodynia to brush | 0-6 hours
Adverse effects | 10 and 30 min after infusion of study medication

CONTACTS AND LOCATIONS:
Overall Officials: Burkhard Gustorff, MD, Study Chair — Medical University of Vienna
Locations (1):
- Department of Anaesthesia, Medical University of Vienna, Vienna, Austria